CLINICAL TRIAL: NCT01458964
Title: Quetiapine Compared With Placebo in the Management of Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Tennessee State University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Norman Moore, Professor, Psychiatry, East Tennessee State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07-032f; NCT00710918 (obsolete NCT alias)
Record Dates: First submitted 2011-10-06; First posted 2011-10-25 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine (Active Comparator): Quetiapine will be administered orally, QHS at a dosage of 100 mg for 1 week increasing to a target dosage of 200 mg for 11 weeks.
  Interventions: Drug: Quetiapine
- Sugar pill (Placebo Comparator): Sugar pill will be administered orally, QHS at a dosage of 100 mg for 1 week increasing to a target dosage of 200 mg for 11 weeks.

INTERVENTIONS:
Drug: Quetiapine — 100 mg (peach colored oblong tablet) and 200 mg (yellow colored oblong tablet)
  Other Names: Seroquel
  Arms: Quetiapine

SUMMARY:
Is quetiapine more effective than other medications in the treatment of fibromyalgia.

DETAILED DESCRIPTION:
This study is a double blind, placebo controlled, 24-week crossover design. For 12 weeks subjects receive either study medication (200mg Quetiapine) or placebo, after which they will be switched to the other treatment for an additional 12 weeks. Between treatments, subjects are required to undergo a 1-week washout where no drug is given in order to clear the effects of the first treatment. At each visit subjects will complete the following assessment: Fibromyalgia Impact Questionnaire, Pittsburgh Sleep Quality Index, Beck Depression Inventory, State-Trait Anxiety Inventory, and Short Form Health Survey. Temperature, blood pressure, pulse rate, weight and waist circumference will also be recorded. Physical exams and blood tests will be performed at 1, 12, and 25 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60, inclusive
* Females of childbearing potential using reliable method of contraception AND negative urine pregnancy test.
* Widespread pain present for at least 3 months
* Widespread encompassing both sides of the body, as well as above and below the waist
* Pain in at least 11 of 18 tender points as determined by a physician

Exclusion Criteria :

* Pregnant or breastfeeding
* Use of any of the following in the 14 days prior to enrollment: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine, saquinavir phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids.
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before enrollment
* Substance or alcohol dependence at enrollment (except in full or recovery, and except nicotine or caffeine dependence)
* Abuse of any of the following within 4 weeks of enrollment: opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen
* Medical conditions that would affect study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomization of treatment in the present study
* Participation in another drug trial within 4 weeks prior to enrollment in this study or longer
* Admitted to hospital for Diabetes Mellitus (DM) related illness in past 12 weeks
* Not under physician's care for DM
* Physician responsible for your DM care has indicated you DM is uncontrolled
* Physician responsible for your DM care has not approved your participation in the study
* Have not been on the same dose of DM medicine and/or diet for the 4 weeks prior to starting the study
* For thiazolidinediones (glitazones) this period should not be less than 8 weeks
* Taking insulin whose daily does on one occasion in the past 4 weeks has been more than 10% above or below your mean dose in the preceding 4 weeks
* A low white blood cell count

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | At 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Norman C Moore, M.D., Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States